CLINICAL TRIAL: NCT03632122
Title: Identifying Subgroups of Older Adults With Back Pain and Multiple Chronic Conditions to Inform Pathways of Care and Improve Population Health
Brief Title: Subgroups of Older Adults With Back Pain and Multiple Chronic Conditions
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Sean Rundell, Assistant Professor, School of Medicine: Rehabilitation Medicine, University of Washington
Other Study IDs: STUDY00005260
Record Dates: First submitted 2018-08-09; First posted 2018-08-15 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Low Back Pain; Depression; Anxiety; Osteoarthritis
Keywords: comorbidity; pain; function; older adults; Medicare
MeSH Terms: conditions — Low Back Pain; Depression; Anxiety Disorders; Osteoarthritis; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bothersome back pain: The investigators will include community-dwelling older adults at Round 1 or 6 of the NHATS cohort, and will include those with bothersome back pain in the past month based on self-report questions at the respective baseline time point. The investigators will exclude participants who are non-ambulatory (requires wheelchair or scooter).

SUMMARY:
The overall goal of this study is to use the National Health and Aging Trends Study (NHATS) data to gain an understanding of how multiple chronic conditions impact the health outcomes of older adults with back pain.

DETAILED DESCRIPTION:
This study seeks to gain knowledge regarding how multiple chronic conditions affect the health and function of older adults with back pain. The investigators will perform a retrospective cohort study using secondary analysis of the National Health and Aging Trends Study (NHATS) data. NHATS collected longitudinal data on Medicare beneficiaries over 65 for six years, from 2011-2017. This set of data is comprehensive and includes self-reported survey data as well as physical performance data, both of which this study will utilize.

The specific aims include to 1) Estimate the longitudinal associations of the number of chronic conditions, using a standard classification scheme, with long-term physical performance, function, and recurrent falls, 2) Identify specific combinations of chronic conditions that are most strongly associated with long-term physical performance, function, and recurrent falls, 3) Determine the association of the number and type of chronic conditions with rehabilitation service use. The investigator will test a corresponding hypothesis for each aim: 1) Medicare beneficiaries reporting back pain with a greater number of chronic conditions will have worse physical performance, lower functional status, and be more likely to experience recurrent falls over 6 years, 2) Medicare beneficiaries reporting back pain with common and potentially modifiable conditions of anxiety, depression, and arthritis (individually and combined as dyads or a triad) will have worse physical performance, lower functional capacity, and be more likely to experience recurrent falls over 6 years, 3) Medicare beneficiaries with back pain and multiple chronic conditions will report lower use of rehabilitation services in the past one year compared to those with back pain alone or one additional chronic condition.

ELIGIBILITY:
Inclusion Criteria:

* This study will include community-dwelling participants in the NHATS study who indicated that in the last month they had been bothered by pain in the last month and indicated that the site of pain was the lower back.

Exclusion Criteria:

* This study will exclude participants who are non-ambulatory (requires wheelchair or scooter).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: NHATS is a cohort of older adults and is representative of Medicare beneficiaries age 65 and older. It is a "unique national resource for the scientific study of functioning in later life." The sample is drawn from the Medicare enrollment files, and the survey oversamples Blacks and those at older ages. Initial NHATS data collection began in 2011 (Round 1) with in-person interviews.
Sampling Method: Probability Sample
Enrollment: 8344 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | 6 years
  NHATS measures physical performance using an in-person physical performance test. The Short Physical Performance Battery, which includes walking 3 meters, balancing activities, and chair stands. Participants are scored from 0 (worst) to 12 (best).
Rehabilitation Use | 1 year
  Participants asked if they had used rehabilitation services over the last year. This is a dichotomous variable of "use" or "no use". If participants answer that they have used rehabilitation services, they are asked the purpose/conditions for which they received care, the body region for which they received care, setting, duration of services in months and weeks, improvement of treatment and whether they met their treatment goals. These are reported as categorical variables.

SECONDARY OUTCOMES:
Walking Capacity | 6 years
  NHATS used survey questions asking about pairs of less or more challenging tasks. This includes walking. The pair of questions corresponding to walking capacity ask participants about their ability to walk 3 and 6 blocks by themselves. Based on their answers participants were put into one of the following categories: unable to do less challenging task able to do less challenging task, able to do less challenging but not more challenging task, able to do the more challenging task. Unable to do less challenging task the least functional capacity and able to do the most challenging task being the highest functional capacity. Higher functional capacity is the better outcome.
Stair Climbing Capacity | 6 years
  NHATS used survey questions asking about pairs of less or more challenging tasks. This includes stair climbing. The pair of questions for stairs asks about the ability to go up 10 and 20 stairs. Based on their answers participants were put into one of the following categories: unable to do less challenging task able to do less challenging task, able to do less challenging but not more challenging task, able to do the more challenging task. Unable to do less challenging task the least functional capacity and able to do the most challenging task being the highest functional capacity. Higher functional capacity is the better outcome.
Falls | 6 years
  The number of "falls" defined as "any fall, slip, or trip in which you lose your balance and land on the floor or ground at a lower level".
Gait Speed | 6 years
  Participants are timed as they finish a three meter walking course.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Rundell SD, Karmarkar A, Nash M, Patel KV. Associations of Multiple Chronic Conditions With Physical Performance and Falls Among Older Adults With Back Pain: A Longitudinal, Population-based Study. Arch Phys Med Rehabil. 2021 Sep;102(9):1708-1716. doi: 10.1016/j.apmr.2021.03.025. Epub 2021 Apr 24. PMID 33901438